CLINICAL TRIAL: NCT01125774
Title: A Six Month Phase II/III, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of Telcagepant (MK-0974) for Prevention of Menstrually Related Migraine in Female Patients With Episodic Migraine
Brief Title: Telcagepant for Prevention of Menstrually Related Migraine in Female Participants With Episodic Migraine (MK-0974-065)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0974-065; 2010_535 (Other: Merck Registration Number)
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Migraine
Keywords: Menstrually related migraine; migraine; Premenstrual migraine
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telcagepant (Experimental): Telcagepant 140 mg was administered once daily at bedtime for 7 consecutive days each month, beginning at the onset of menses, for up to 6 months. Dosing could begin up to 3 days prior to menses onset if prodromal symptoms reliably predicted onset of menses.
  Interventions: Drug: Telcagepant
- Placebo (Placebo Comparator): Placebo was administered once daily at bedtime for 7 consecutive days each month, beginning at the onset of menses, for up to 6 months. Dosing could begin up to 3 days prior to menses onset if prodromal symptoms reliably predicted onset of menses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telcagepant — Telcagepant 140 mg film coated tablet for oral administration
  Other Names: MK-0974
  Arms: Telcagepant
Drug: Placebo — Placebo to match telcagepant 140 mg film coated tablet for oral administration
  Arms: Placebo

SUMMARY:
This is a multicenter study to test the hypothesis that telcagepant is superior to placebo in preventing perimenstrual migraines as measured by mean monthly headaches during the entire treatment period. This study will also evaluate the safety and tolerability of telcagepant for female migraine participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant who has had regular menstrual cycles monthly (22 to 32 days) for at least the last 3 cycles
* Participant experiences headache during menstrual period in at least 2 out of last 3 cycles
* Participant has history of migraine for ≥ 3 months and with ≥ 2 migraine attacks per month in the 2 months prior to screening
* Participant agrees to use an effective method of birth control through the duration of the study

Exclusion Criteria:

* Participant has basilar or hemiplegic migraine headache
* Participant has taken medication for acute headache on more than 15 days per month in the 3 months prior to screening
* Participant is taking prophylactic medication for migraine and daily dose has changed within 4 weeks prior to screening
* Participant has history of significant liver disease
* Participant has had cardiac surgery or symptoms within 3 months of screening
* Participant has confounding pain syndromes, psychiatric conditions, dementia, or major neurological disorders other than migraine
* Participant has history of neoplastic disease ≤ 5 years prior to signing informed consent
* Participant has history of gastric or small intestinal surgery
* Participant consumes 3 or more alcoholic drinks per day

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4548 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2011-04-08 (Actual); Study Completion 2011-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Ho TW, Ho AP, Ge YJ, Assaid C, Gottwald R, MacGregor EA, Mannix LK, van Oosterhout WP, Koppenhaver J, Lines C, Ferrari MD, Michelson D. Randomized controlled trial of the CGRP receptor antagonist telcagepant for prevention of headache in women with perimenstrual migraine. Cephalalgia. 2016 Feb;36(2):148-61. doi: 10.1177/0333102415584308. Epub 2015 Apr 29. PMID 25926620
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-065&kw=0974-065&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to telcagepant 140 mg or placebo. Protocol deviation occurred in which 28 participants (called "duplicate participants") were randomized at more than 1 study site (22 unique participants randomized in total 37 times to telcagepant and 12 times to placebo; 6 unique participants randomized in total 12 times to placebo)
Groups:
- Telcagepant 140 mg - Excluding Duplicate Participants: Participants who were randomized at only 1 study site and were randomized to telcagepant. Telcagepant 140 mg was administered once daily at bedtime for 7 consecutive days each month, beginning at the onset of menses, for up to 6 months. Dosing could begin up to 3 days prior to menses onset if prodromal symptoms reliably predicted onset of menses.
- Placebo - Excluding Duplicate Participants: Participants who were randomized at only 1 study site and were randomized to placebo. Placebo was administered once daily at bedtime for 7 consecutive days each month, beginning at the onset of menses, for up to 6 months. Dosing could begin up to 3 days prior to menses onset if prodromal symptoms reliably predicted onset of menses.
- Telcagepant 140 mg - Duplicate Participants: Participants who were randomized at more than 1 study site and were randomized at least once to telcagepant and may also have been randomized to placebo. Study drug was administered once daily at bedtime for 7 consecutive days each month, beginning at the onset of menses, for up to 6 months. Dosing could begin up to 3 days prior to menses onset if prodromal symptoms reliably predicted onset of menses.
- Placebo - Duplicate Participants: Participants who were randomized at more than 1 study site and each time were randomized to placebo. Placebo was administered once daily at bedtime for 7 consecutive days each month, beginning at the onset of menses, for up to 6 months. Dosing could begin up to 3 days prior to menses onset if prodromal symptoms reliably predicted onset of menses.
Period: Overall Study
Arm/Group | Telcagepant 140 mg - Excluding Duplicate Participants | Placebo - Excluding Duplicate Participants | Telcagepant 140 mg - Duplicate Participants | Placebo - Duplicate Participants
Started | 3018 (Randomized) | 1502 (Randomized) | 22 (Unique participants randomized) | 6 (Unique participants randomized)
Treated | 2638 | 1322 (1 mistakenly took telcagepant and is included with telcagepant group for adverse event analysis) | 21 (Received telcagepant) | 5
Completed | 1893 | 948 | 13 (Completed study at least once while treated with telcagepant (otherwise counted "Not Completed")) | 3 (Completed study at least once)
Not Completed | 1125 | 554 | 9 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants, including those randomized at more than 1 site ("duplicate participants"). Participants randomized at more than 1 site resulting in randomization into both telcagepant 140 mg and placebo groups are allocated to the telcagepant 140 mg group.
Groups:
- Telcagepant 140 mg: Telcagepant 140 mg was administered once daily at bedtime for 7 consecutive days each month, beginning at the onset of menses, for up to 6 months. Dosing could begin up to 3 days prior to menses onset if prodromal symptoms reliably predicted onset of menses.
- Total: Total of all reporting groups
Arm/Group | Telcagepant 140 mg | Placebo | Total
Number analyzed (Participants) | 3040 | 1508 | 4548
Age, Continuous [Mean (Standard Deviation); unit: Years] — Due to missing data, N=3039 and 4547 for Telcagepant 140 mg and Total groups, respectively.
  Years | 36.1 (8.6) | 35.8 (8.7) | 36.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3040 | 1508 | 4548
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Adverse Events (AEs)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study drug, is also an AE. A clinical AE is an AE reported as a result of a clinical examination or reported by the participant.
Time Frame: Up to 14 days after the last dose of study drug (Up to 6.5 months)
Population: All Participants as Treated (APaT) population, which included all randomized participants who took at least one dose of study drug. Participants were included in the treatment arm corresponding to the study treatment actually taken. Participants who took both study treatments were included in the telcagepant 140 mg treatment arm.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 2660 | 1326
Participants | 1582 (0.19) | 804 (0.26)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; Miettinen & Nurminen; Difference in percent incidence = -1.2, 95% CI 2-sided [-4.4 to 2.1] — Telcagepant percent incidence versus Placebo percent incidence

2. Primary Outcome: Number of Participants Who Discontinued Study Due to a Clinical AE
Description: as for outcome 1
Time Frame: Up to 6 months
Population: APaT population, which included all randomized participants who took at least one dose of study drug. Participants were included in the treatment arm corresponding to the study treatment actually taken. Participants who took both study treatments were included in the telcagepant 140 mg treatment arm.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 2660 | 1326
Participants | 66 (0.19) | 36 (0.26)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; Miettinen & Nurminen; Difference in percent incidence = -0.2, 95% CI 2-sided [-1.4 to 0.8] — Telcagepant percent incidence versus Placebo percent incidence

3. Primary Outcome: Number of Participants With Laboratory AEs
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the study drug, is also an AE. A laboratory AE is an AE reported as a result of a laboratory assessment or test.
Time Frame: Up to 6 months
Population: APaT population, which is all randomized participants who took at least one dose of study drug. Also to be included participant must have at least one post-baseline lab test. Participants were included in arm corresponding to the treatment actually taken. Participants who took both treatments were included in the telcagepant 140 mg treatment arm.
Measure: Number; unit: Participants
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 2610 | 1305
Participants | 76 (0.19) | 30 (0.26)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; Miettinen & Nurminen; Difference in percent incidence = 0.6, 95% CI 2-sided [-0.5 to 1.6] — Telcagepant percent incidence versus Placebo percent incidence

4. Primary Outcome: Number of Participants Who Discontinued Study Due to a Laboratory AE
Description: as for outcome 3
Time Frame: Up to 6 months
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 2610 | 1305
Participants | 8 (0.19) | 2 (0.26)

5. Primary Outcome: Mean Monthly Headache Days During Entire Study Period Among Participants With Menstrually-related Migraine (MRM) or Pure Menstrual Migraine (PMM) Who Have an Average of 5 or More Moderate or Severe Migraine Headaches Per Month at Baseline
Description: Participants completed a headache diary each evening at bedtime, including recording headache duration and acute headache medication use. Mean monthly headache days was calculated from diary data. A headache day was defined as a day in which a headache (defined as headache pain ≥30 minute duration or requiring acute treatment) started, ended, or recurred. Headache pain persisting for more than 1 calendar day after initial onset was considered an occurrence of additional headache days. Mean monthly rate was adjusted to 28 days. Participant subgroups (based on symptoms over the 3 menstrual cycles prior to study): PMM - In ≥2 out of 3 cycles attacks occur exclusively on Day 1 ± 2 of menstruation and at no other times of the cycle; MRM - In ≥2 out of 3 cycles attacks occur on Day 1 ± 2 of menstruation and additionally at other times of the cycle.
Time Frame: Up to 6 months
Population: All randomized participants who were randomized only once, took at least 1 dose of study drug, had ≥1 post-randomization efficacy measurement, met the definition of the MRM or PMM subgroup and reported average of ≥5 moderate-severe migraine headaches/month at baseline. Participant must have ≥1 month with ≥4 dosing days and ≥7 diary days.
Measure: Mean (Standard Error); unit: Days per month
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 887 | 447
Days per month | 8.8 (0.19) | 9.3 (0.26)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; This measure tests the primary hypothesis, that telcagepant 140 mg is superior to placebo as measured by mean monthly headache days in participants with MRM or PMM; Test type: Superiority or Other; p = 0.130, Longitudinal data analysis (LDA) — α=0.0499; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.1] — Difference is Telcagepant 140 mg versus Placebo

6. Secondary Outcome: Mean Monthly Headache Days During Entire Study Period Among Participants With MRM Who Have an Average of 5 or More Moderate or Severe Migraine Headaches Per Month at Baseline
Description: Participants completed a headache diary each evening at bedtime, including recording headache duration and acute headache medication use. Mean monthly headache days was calculated from diary data. A headache day was defined as a day in which a headache (defined as headache pain ≥30 minute duration or requiring acute treatment) started, ended, or recurred. Headache pain persisting for more than 1 calendar day after initial onset was considered an occurrence of additional headache days. Mean monthly rate was adjusted to 28 days. MRM participant subgroup (based on symptoms over the 3 menstrual cycles prior to study) - In ≥2 out of 3 cycles attacks occur on Day 1 ± 2 of menstruation and additionally at other times of the cycle.
Time Frame: Up to 6 months
Population: All randomized participants who were randomized only once, took at least 1 dose of study drug, had ≥1 post-randomization efficacy measurement, met the definition of the MRM subgroup and reported average of ≥5 moderate-severe migraine headaches/month at baseline. Participant must have ≥1 month with ≥4 dosing days and ≥7 diary days.
Measure: Mean (Standard Error); unit: Days per month
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 731 | 382
Days per month | 9.3 (0.20) | 9.6 (0.28)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p = 0.369, LDA — To control Type I error, formal significance of the test for treatment difference for this measure could only be achieved if the comparison corresponding to the primary hypothesis was significant at α=0.0499; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.4] — Difference is Telcagepant 140 mg versus Placebo

7. Secondary Outcome: Mean Monthly On-drug Headache Days During the Entire Study Period Among Participants With MRM or PMM Who Have an Average of 5 or More Moderate or Severe Migraine Headaches Per Month at Baseline
Description: Participants completed a headache diary each evening at bedtime, including recording headache duration and acute headache medication use. Mean monthly on-drug headache days was calculated from diary data. "On-drug" headache day was a day, which had a valid diary entry and which followed a study drug dosing day, in which a headache (defined as headache pain ≥30 minute duration or requiring acute treatment) started, ended, or recurred. Headache pain persisting for more than 1 calendar day after initial onset into additional qualifying days (i.e., day following dosing day) was considered an occurrence of additional headache days. Mean monthly rate was adjusted to 7 days. Participant subgroups (based on symptoms over the 3 menstrual cycles prior to study): PMM - In ≥2 out of 3 cycles attacks occur exclusively on Day 1 ± 2 of menstruation and at no other times of the cycle; MRM - In ≥2 out of 3 cycles attacks occur on Day 1 ± 2 of menstruation and additionally at other times of the cycle.
Time Frame: Up to 6 months
Population: All randomized participants who were randomized only once, took at least 1 dose of study drug, had ≥1 post-randomization efficacy measurement, met the definition of the MRM or PMM subgroup and reported average of ≥5 moderate-severe migraine headaches/month at baseline. Participant must have ≥1 month with ≥4 dosing days.
Measure: Mean (Standard Error); unit: Days per month
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 887 | 448
Days per month | 2.5 (0.05) | 2.9 (0.08)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, LDA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.5 to -0.2] — Difference is Telcagepant 140 mg versus Placebo

8. Secondary Outcome: Mean Monthly On-drug Headache Days During the Entire Study Period Among Participants With MRM Who Have an Average of 5 or More Moderate or Severe Migraine Headaches Per Month at Baseline
Description: Participants completed a headache diary each evening at bedtime, including recording headache duration and acute headache medication use. Mean monthly on-drug headache days was calculated from diary data. "On-drug" headache day was a day, which had a valid diary entry and which followed a study drug dosing day, in which a headache (defined as headache pain ≥30 minute duration or requiring acute treatment) started, ended, or recurred. Headache pain persisting for more than 1 calendar day after initial onset into additional qualifying days (i.e., day following dosing day) was considered an occurrence of additional headache days. Mean monthly rate was adjusted to 7 days. MRM participant subgroup (based on symptoms over the 3 menstrual cycles prior to study) - In ≥2 out of 3 cycles attacks occur on Day 1 ± 2 of menstruation additionally at other times of the cycle.
Time Frame: Up to 6 months
Population: All randomized participants who were randomized only once, took at least 1 dose of study drug, had ≥1 post-randomization efficacy measurement, met the definition of the MRM subgroup and reported average of ≥5 moderate-severe migraine headaches/month at baseline. Participant must have ≥1 month with ≥4 dosing days.
Measure: Mean (Standard Error); unit: Days per month
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 731 | 383
Days per month | 2.6 (0.06) | 3.0 (0.08)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p < 0.001, LDA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.2] — Difference is Telcagepant 140 mg versus Placebo

9. Secondary Outcome: Mean Monthly On-drug Headache Days During the Entire Study Period Among Participants With PMM Who Have an Average of 3 or More Moderate or Severe Migraine Headaches Per Month at Baseline
Description: Participants completed a headache diary each evening at bedtime, including recording headache duration and acute headache medication use. Mean monthly on-drug headache days was calculated from diary data. "On-drug" headache day was a day, which had a valid diary entry and which followed a study drug dosing day, in which a headache (defined as headache pain ≥30 minute duration or requiring acute treatment) started, ended, or recurred. Headache pain persisting for more than 1 calendar day after initial onset into additional qualifying days (i.e., day following dosing day) was considered an occurrence of additional headache days. Mean monthly rate was adjusted to 7 days. PMM participant subgroups (based on symptoms over the 3 menstrual cycles prior to study) - In ≥2 out of 3 cycles attacks occur exclusively on Day 1 ± 2 of menstruation and at no other times of the cycle.
Time Frame: Up to 6 months
Population: All randomized participants who were randomized only once, took at least 1 dose of study drug, had ≥1 post-randomization efficacy measurement, met the definition of the PMM subgroup and reported average of ≥3 moderate-severe migraine headaches/month at baseline. Participant must have ≥1 month with ≥4 dosing days.
Measure: Mean (Standard Error); unit: Days per month
Arm/Group | Telcagepant 140 mg | Placebo
Number analyzed (Participants) | 344 | 151
Days per month | 2.1 (0.08) | 2.2 (0.12)
Statistical Analysis 1: Comparison: Telcagepant 140 mg vs Placebo; Test type: Superiority or Other; p = 0.393, LDA — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.4 to 0.2] — Difference is Telcagepant 140 mg versus Placebo

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose of study drug (Up to 6.5 months)
Description: APaT population, which included all randomized participants who took at least 1 dose of study drug. Participants were included in the treatment arm corresponding to the study treatment actually taken. Participants who took both study treatments were included in the telcagepant 140 mg treatment arm. Presentation includes clinical and laboratory AEs.
Arm/Group | Telcagepant 140 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 25/2660 | 10/1326
Other Adverse Events (participants affected / at risk) | 819/2660 | 413/1326
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telcagepant 140 mg (N=2660) | Placebo (N=1326)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cervicitis (Infections and infestations) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telcagepant 140 mg (N=2660) | Placebo (N=1326)
Diarrhoea (Gastrointestinal disorders) | 186 (292) | 90 (128)
Dry mouth (Gastrointestinal disorders) | 174 (359) | 85 (168)
Nausea (Gastrointestinal disorders) | 270 (467) | 165 (264)
Fatigue (General disorders) | 135 (194) | 65 (130)
Nasopharyngitis (Infections and infestations) | 190 (226) | 102 (122)
Dizziness (Nervous system disorders) | 204 (340) | 100 (166)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.